CLINICAL TRIAL: NCT06951321
Title: Clinical and Pathophysiological Characteristics of Postinfectious Cough Post COVID-19 Infection: a Multi-center Nationwide Research
Brief Title: Characteristics of Postinfectious Cough
Status: Completed | Type: Observational
Sponsor: Kefang Lai (Other)
Responsible Party: Sponsor-Investigator, Kefang Lai, professor, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: ES-2023-032-01
Record Dates: First submitted 2025-04-14; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cough
Keywords: cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples (200 cases), sputum supernatant (200 cases), original sputum (200 cases)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients

SUMMARY:
Collect the age, sex and other demographic data of 1600 patients with chronic cough after COVID-19 infection and clinical parameters such as cough characteristics, establish a cohort of patients with chronic cough after COVID-19 infection, observe the type and level of airway inflammation, airway responsiveness, cough sensitivity and changes in microbiology of patients with chronic cough after COVID-19 infection, clarify the epidemiological characteristics, clinical pathophysiological characteristics, long-term prognosis and related factors of patients with chronic cough after COVID-19 infection, explore the clinical pathophysiological characteristics and pathogenesis of cough after COVID-19 infection, and provide a theoretical basis for the treatment of persistent cough after COVID-19 infection.

DETAILED DESCRIPTION:
1. Formulate clinical data registration questionnaire (including baseline and follow-up) Adopt the form of online questionnaire survey, unify the inclusion criteria, and register the demographic characteristics of patients with cough after COVID-19 infection and the clinical data of acute infection and migration, including the symptoms of COVID-19 infection in the acute phase, the characteristics related to the current cough symptoms (such as cough phase, nature, severity assessment, etc.), past disease history, current drug use, etc. It is expected that there will be no less than 1600 postinfecitous cough questionnaires. Simultaneously record the laboratory test results of the patient, including blood cell classification count, lung ventilation and bronchial provocation test, induced sputum analysis, fractional exhaled nitric oxide , chest X-ray or CT examination, sputum bacterial culture (for cough patients), besides, some patients have completed cough stimulation tests. Secondly, follow-up visits (12 weeks, 52 weeks) were conducted on the included postinfectious cough patients to record the characteristics and severity of cough symptoms in the delayed patients. Some patients were re-examined for lung ventilation and bronchial provocation tests, cough provocation tests, induced sputum analysis, and fractional exhaled nitric oxide, and the results were recorded. Among them, serum samples (200 cases), sputum supernatant (200 cases), and original sputum (200 cases) were collected.
2. Analysis of airway microbiome in postinfectious cough post COVID-19 patients The patients with cough after COVID-19 infection and the healthy subjects matched in age and sex were included. The original sputum was obtained for macro gene sequencing. In addition, the sputum supernatant and sputum cells were separated by induced sputum treatment. The sputum supernatant was used for metabolic group and inflammatory factor detection, the sputum cells were used for transcriptome sequencing, the Illumina HiSeq2500 was used for macro genome and transcriptome sequencing, LC-MS/MS was used for non targeted metabolic group detection, and Luminex multi factor kit was used for inflammatory factor detection. Through dimensional reduction analysis of the obtained multiomics data, a multivariable linear mixed model was established, and clinical indicators were used as covariates to carry out association analysis of the multiomics data, in order to identify the key genes of the cross integration of multiomics biological pathway and the species encoding the gene, and to obtain the "flora metabolism host inflammation" pathway that significantly interacts in the cough after COVID-19 infection, thereby revealing the potential mechanism of COVID-19 infection induced cough persistence.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-70 years old, gender not limited;
2. After COVID-19 infection (COVID-19 nucleic acid test or antigen test is positive, or there is a highly suspected symptom of COVID-19 infection), the cough lasts for more than 3 weeks and there is still cough at the time of investigation;
3. No obvious abnormalities were found in chest imaging.

Exclusion Criteria:

1. Combined with other respiratory infectious diseases (pneumonia, tuberculosis, etc.);
2. Combined chronic respiratory diseases (asthma, chronic obstructive pulmonary disease, bronchiectasis, interstitial lung disease, etc.);
3. Cough and expectoration were found 2 months before COVID-19 infection;
4. Merge other serious organ diseases and malignant tumors;
5. Pregnant and lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cough lasts for more than 3 weeks after COVID-19 infection and there is still cough at the time of investigation
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
cough duration | From enrollment to 1 year after the enrollment
  The total cough duration after COVID-19 infection reported by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Considering that patients are unwilling to disclose their personal privacy information. If necessary, please contact us and we will consider providing it.